CLINICAL TRIAL: NCT05126693
Title: Algorithms for Patient-specific Treatment Planning in Cerebral Palsy Based on the Muscle and Tendon Architecture - Short Term Follow-up of a Botulinum Toxin Intervention in Children With Spastic Cerebral Palsy
Brief Title: Short Term Follow-up of a Botulinum Toxin Intervention in Children With Spastic Cerebral Palsy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Collaborators: KU Leuven (Other)
Responsible Party: Principal Investigator, Kaat Desloovere, Prof. Dr., Universitaire Ziekenhuizen KU Leuven
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: S59945_C
Record Dates: First submitted 2021-08-17; First posted 2021-11-19 (Actual); Results first posted 2025-07-31 (Actual); Last update posted 2025-07-31 (Actual); Status verified 2025-05

CONDITIONS: Spastic Cerebral Palsy
Keywords: Cerebral Palsy; Spastic Cerebral Palsy; Botulinum Toxin; muscle morphology; Range of motion; Stiffness; Spasticity; Intensive physical therapy
MeSH Terms: conditions — Cerebral Palsy; Muscle Spasticity

STUDY DESIGN:
Intervention Model Description: We will include patients who receive BoNT injections at the lower limb in the intervention group. Patient with no indication for treatment in the next three months (besides the routine physical therapy and orthotic management) will be asked to participate in the control group. Justification for the non-randomized design is stated above.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): The children in the intervention group will receive BoNT injections in the medial gastrocnemius and/or the semitendinosus muscle(s). As part of the standard treatment approach of the CP Reference Centre of the University Hospitals Leuven, the injections are followed by a period of bilateral stretching casts if indicated (below the knee walking casts and removable knee extension casts when necessary) and all children will receive intensive physical therapy and application of ankle foot orthoses following BoNT injections. The follow-up period for the current study is 8-10 weeks. During this intensive physical therapy period post-BoNT, the children in the intervention group will work on individualized treatment goals, which will be defined based on the baseline measurements during a multidisciplinary discussion with the treating physician (that is scheduled prior to the BoNT injections).
  Interventions: Other: Botulinum Toxin treatment combined with a post-BoNT intensive physical therapy period guided by individualized treatment goals.
- Control group (No Intervention): This group will continue their usual care or normal routine treatment, i.e. physiotherapy and orthotic management during a period of 8-10 weeks.

INTERVENTIONS:
Other: Botulinum Toxin treatment combined with a post-BoNT intensive physical therapy period guided by individualized treatment goals. — BoNT treatment combined with a follow-up period of intensive physical therapy of 8-10 weeks. During this intensive physical therapy post BoNT injections, the children in the intervention group will work on individualized treatment goals, which will be defined based on the baseline measurements during a multidisciplinary discussion with the treating physician (planned prior to the BoNT injections).
  Arms: Intervention group

SUMMARY:
This study investigates the effect of integrated Botulinum Neurotoxin A (BoNT) treatment on morphologic muscle and tendon properties, spasticity, joint stiffness, joint range of motion, muscle strength, gait and gross motor function. The integrated BoNT treatment combines BoNT-injections with serial casting and intensive physical therapy, as previously described by Molenaers et al. The current study will include 30 children who are clinically scheduled for BoNT treatment in the medial gastrocnemius and/or the semitendinosus muscle in the intervention group and 30 children in a control group who will receive usual care within a time span of 3 months.

DETAILED DESCRIPTION:
Aim:

This study investigates the effect of integrated Botulinum Neurotoxin A (BoNT) treatment on morphologic muscle and tendon properties (muscle length and muscle volume, assessed with a 3D ultrasound measurement), spasticity and joint stiffness (measured with an instrumented spasticity assessment), joint range of motion (measured through goniometry), muscle strength (measured using dynamometry), gait (assessed through 3D gait analysis) and gross motor function (assessed using clinical test batteries). The aim is twofold: (1) determine whether integrated BoNT treatment of the medial gastrocnemius and the semitendinosus muscle(s) leads to changes in the morphologic muscle and tendon properties of the medial gastrocnemius and the semitendinosus muscle(s), the ankle and knee range of motion, spasticity, stiffness, muscle strength and gait, and (2) determine the correlation between baseline morphologic muscle and tendon properties and the changes in the primary outcome parameters (spasticity and stiffness) following the BoNT-treatment.

Design:

The current study has a non-randomized controlled design. Because BoNT is proven an effective treatment to reduce spasticity and improve gross motor function, it cannot be clinically justified to allocate children to a non-treatment group, if a new BoNT treatment is required. Delayed BoNT treatment could rapidly increase musculoskeletal impairments. It is therefore considered unethical to temporarily withdraw BoNT treatment from patients. To compensate the lack of randomization accurate matching of groups is required. Children will be matched on diagnosis (uni/bilateral CP), GMFCS level, age and spasticity level.

BoNT-treatment:

All children in the intervention group will receive BoNT injections in the medial gastrocnemius and/or the semitendinosus muscle(s) (other muscles may also be treated as part of multilevel treatment). As part of the standard integrated treatment approach of the CP Reference Centre of the University Hospitals Leuven, the injections are followed by a period of bilateral stretching casts if indicated (below the knee walking casts and removable knee extension casts when necessary) and all children will receive intensive physical therapy and application of orthotic management following BoNT injections. The follow-up period for the current study is 8-10 weeks. During this intensive physical therapy post-BoNT, the children in the intervention group will work on individualized treatment goals. These goals will be defined based on the baseline measurements during a multidisciplinary discussion with the treating physician, which is scheduled prior to the BoNT treatment. The fulfillment of these patient-specific goals will be evaluated by the Goal Attainment Score (GAS). During the follow-up period, the treating physical therapist will be interviewed on a two-weekly basis to verify whether and to what extend the therapy is focused on the personal treatment goals. Assessments of morphologic muscle and tendon properties, spasticity, stiffness, joint range of motion, muscle strength, and gait of the participants will be performed before the BoNT injections, and 8-10 weeks after the injection. This period of 8-10 weeks follow-up post BoNT injections was found to be appropriate, since the potential effect of BoNT on gross motor function is expected to be optimal after 6-10 weeks.

Study groups:

The study will include patients who are diagnosed with spastic CP, aged between 4 and 11 years and with Gross Motor Function Classification System (GMFCS) level I-III. The intervention and control group will be group-matched based on diagnosis (uni/lateral CP), GMFCS level, age and spasticity level.

Overall exclusion criteria were: BoNT injections less than 6 months before inclusion, a treatment history that includes previous selective dorsal rhizotomy treatment or a bony surgery less than 2 years before inclusion, and limited cooperation that would prevent a proper assessment. For all enrolled children, intensive rehabilitation post BoNT injections had to be foreseen as the standard care. For the intervention group, 30 children with a clinical indication for BoNT injections in the medial gastrocnemius and/or semitendinosus muscle(s) will be recruited, while for the control group, 30 children without an indication for a specific intervention in the next 3 months will be recruited.

For the intervention group, the baseline measures will be followed by the BoNT injections combined with casting and goal-oriented physical therapy (as described above), and the follow-up assessments will be planned 8-10 weeks post BoNT injections. Baseline and follow-up assessments for the intervention groups include 3D ultrasound, the instrumented spasticity measurement, functional strength tests, and 3D gait analysis.

The children in the control group will also be assessed twice with an interval of 8-10 weeks. During the 8-10 weeks, they will continue their usual care or normal routine treatment, i.e. regular physiotherapy and orthotic devices. Baseline and follow-up assessments for the control group include 3D ultrasound, the instrumented spasticity measurement and functional strength tests.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of spastic cerebral palsy
* Aged 4-11 years
* GMFCS levels I-III (GMFCS = Gross Motor Function Classification Score, expressing the overall functional level of impairment)
* Sufficient cooperation to comprehend and complete the test procedure
* Additional exclusion criterion for the intervention group specifically: Indication for BoNT injections

Exclusion Criteria:

* Non-ambulatory
* Botulinum toxin A injections six months prior to enrollment
* Lower limb surgery two years prior to enrollment
* Previous selective dorsal rhizotomy
* Presence of ataxia or dystonia
* Cognitive problems that impede measurements
* Severe co-morbidities (severe epilepsy, non-correctable visual impairment, autism spectrum disorders, mental problems that prevent comprehensiveness of the tasks)
* Hospitalization after the BoNT treatment for intensive physical therapy
* Intrathecal baclofen pump
* For the control group: new intervention planned within 3 months
* Additional exclusion criterion for the control group specifically: new intervention planned within 3 months

Ages: 4 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 61 (Actual)
Dates: Start 2020-08-03 (Actual); Primary Completion 2022-05-10 (Actual); Study Completion 2022-05-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kaat Desloovere, Prof. Dr., Principal Investigator — UZ Leuven
Locations (1):
- UZ Leuven, Leuven, Vlaams-Brabant, Belgium

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Bar-On L, Aertbelien E, Molenaers G, Van Campenhout A, Vandendoorent B, Nieuwenhuys A, Jaspers E, Hunaerts C, Desloovere K. Instrumented assessment of the effect of Botulinum Toxin-A in the medial hamstrings in children with cerebral palsy. Gait Posture. 2014 Jan;39(1):17-22. doi: 10.1016/j.gaitpost.2013.05.018. Epub 2013 Jun 20. PMID 23791154
- [Background] Bar-On L, Van Campenhout A, Desloovere K, Aertbelien E, Huenaerts C, Vandendoorent B, Nieuwenhuys A, Molenaers G. Is an instrumented spasticity assessment an improvement over clinical spasticity scales in assessing and predicting the response to integrated botulinum toxin type a treatment in children with cerebral palsy? Arch Phys Med Rehabil. 2014 Mar;95(3):515-23. doi: 10.1016/j.apmr.2013.08.010. Epub 2013 Aug 27. PMID 23994052
- [Background] Franki I, Bar-On L, Molenaers G, Van Campenhout A, Craenen K, Desloovere K, Feys H, Pauwels P, De Cat J, Ortibus E. Tone Reduction and Physical Therapy: Strengthening Partners in Treatment of Children with Spastic Cerebral Palsy. Neuropediatrics. 2020 Apr;51(2):89-104. doi: 10.1055/s-0039-3400987. Epub 2019 Nov 27. PMID 31777043
- [Background] Franki I, Desloovere K, De Cat J, Feys H, Molenaers G, Calders P, Vanderstraeten G, Himpens E, Van Broeck C. The evidence-base for basic physical therapy techniques targeting lower limb function in children with cerebral palsy: a systematic review using the International Classification of Functioning, Disability and Health as a conceptual framework. J Rehabil Med. 2012 May;44(5):385-95. doi: 10.2340/16501977-0983. PMID 22549646
- [Background] Molenaers G, Fagard K, Van Campenhout A, Desloovere K. Botulinum toxin A treatment of the lower extremities in children with cerebral palsy. J Child Orthop. 2013 Nov;7(5):383-7. doi: 10.1007/s11832-013-0511-x. Epub 2013 Aug 28. PMID 24432099
- [Background] Peeters N, Van Campenhout A, Hanssen B, Cenni F, Schless SH, Van den Broeck C, Desloovere K, Bar-On L. Joint and Muscle Assessments of the Separate Effects of Botulinum NeuroToxin-A and Lower-Leg Casting in Children With Cerebral Palsy. Front Neurol. 2020 Apr 21;11:210. doi: 10.3389/fneur.2020.00210. eCollection 2020. PMID 32373040
- [Background] Cenni F, Monari D, Desloovere K, Aertbelien E, Schless SH, Bruyninckx H. The reliability and validity of a clinical 3D freehand ultrasound system. Comput Methods Programs Biomed. 2016 Nov;136:179-87. doi: 10.1016/j.cmpb.2016.09.001. Epub 2016 Sep 6. PMID 27686714
- [Background] Bar-On L, Aertbelien E, Wambacq H, Severijns D, Lambrecht K, Dan B, Huenaerts C, Bruyninckx H, Janssens L, Van Gestel L, Jaspers E, Molenaers G, Desloovere K. A clinical measurement to quantify spasticity in children with cerebral palsy by integration of multidimensional signals. Gait Posture. 2013 May;38(1):141-7. doi: 10.1016/j.gaitpost.2012.11.003. Epub 2012 Dec 4. PMID 23218728
- [Background] Molenaers, G., Desloovere, K., Eyssen, M., Decaf, J., Jonkers, I., & Cock, P. De. (1999). Botulinum toxin type A treatment of cerebral palsy: an integrated approach. European Journal of Neurology, 6, s51-s57. https://doi.org/10.1111/j.1468-1331.1999.tb00035.x
- [Result] Peeters N, Papageorgiou E, Hanssen B, De Beukelaer N, Staut L, Degelaen M, Van den Broeck C, Calders P, Feys H, Van Campenhout A, Desloovere K. The Short-Term Impact of Botulinum Neurotoxin-A on Muscle Morphology and Gait in Children with Spastic Cerebral Palsy. Toxins (Basel). 2022 Sep 29;14(10):676. doi: 10.3390/toxins14100676. PMID 36287944
- [Result] Peeters N, Hanssen B, Bar-On L, De Groote F, De Beukelaer N, Coremans M, Van den Broeck C, Dan B, Van Campenhout A, Desloovere K. Associations between muscle morphology and spasticity in children with spastic cerebral palsy. Eur J Paediatr Neurol. 2023 May;44:1-8. doi: 10.1016/j.ejpn.2023.01.007. Epub 2023 Jan 10. PMID 36706682

RESULTS

PARTICIPANT FLOW:
Groups:
- Intervention Group: The children in the intervention group will receive BoNT injections in the medial gastrocnemius and/or the semitendinosus muscle(s). As part of the standard treatment approach of the CP Reference Centre of the University Hospitals Leuven, the injections are followed by a period of bilateral stretching casts if indicated (below the knee walking casts and removable knee extension casts when necessary).
  All children will then undergo an intensive physical therapy program lasting 8-10 weeks. This post-BoNT therapy phase is guided by individualized treatment goals, which are established based on baseline assessments. These goals are determined during a multidisciplinary meeting with the treating physician, held prior to the BoNT injections.
  Thus, the intervention consists of BoNT treatment combined with an 8-10 week period of intensive physical therapy tailored to each child's specific therapeutic needs.
Period: Pre-BoNT/ Pre-3DfUS
Arm/Group | Intervention Group | Control Group
Started | 31 | 30
Completed | 25 | 20
Not Completed | 6 | 10
Not completed — Bad 3DGA data | 2 | 0
Not completed — No 3DGA | 4 | 0
Not completed — Insufficient matching | 0 | 10
Period: 8-10w Post-BoNT/ 8-10w Post-3DfUS
Arm/Group | Intervention Group | Control Group
Started | 25 | 20
Completed | 25 | 20
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intervention Group | Control Group | Total
Number analyzed (Participants) | 25 | 20 | 45
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 25 | 20 | 45
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Median (Inter-Quartile Range); unit: Years] | 6.4 [4.6 to 8.5] | 7.6 [6.2 to 9.4] | 7.1 [5.9 to 9.1]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 4 | 16
  Male | 13 | 16 | 29
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Belgium | 25 | 20 | 45

OUTCOME MEASURES:

1. Primary Outcome: Change in Normalized Muscle Volume of the Medial Gastrocnemius and the Distal Compartment of the Semitendinosus
Description: Estimation of the muscle belly volume by three-dimensional freehand ultrasonography normalized to the product of body weight and height
Time Frame: Between baseline and 8-10 weeks after the BoNT injections for the intervention group, and between baseline and 8-10 weeks later for the control group.
Population: Semitendinosus:
  Intervention group: n = 24 < 25 due to bad quality data Control group: n = 19 < 20 due to bad quality data
Measure: Median (Inter-Quartile Range); unit: ml/kg*m
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 25 | 20
ml/kg*m
  Medial Gastrocnemius | -0.08 [-0.16 to 0.04] | 0.00 [-0.09 to 0.06]
  Semitendinosus: number analyzed (Participants) | 24 | 19
  Semitendinosus | -0.09 [-0.16 to 0.01] | -0.01 [-0.07 to 0.04]

2. Primary Outcome: Change in Echogenicity Intensity of the Medial Gastrocnemius and the Distal Compartment of the Semitendinosus
Description: Estimation of the echogenicity intensity of the whole muscle volume by three-dimensional freehand ultrasonography. Echogenicity is expressed in arbitrary units ranging from 0 to 255. Higher values indicate lighter images, which indirectly suggests the presence of more non-contractile muscle tissue.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: Arbitrary units ranging from 0 to 255
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 25 | 20
Arbitrary units ranging from 0 to 255
  Medial Gastrocnemius | 2.74 [-5.63 to 11.11] | -0.08 [-3.77 to 9.33]
  Semitendinosus: number analyzed (Participants) | 24 | 19
  Semitendinosus | 6.58 [-8.27 to 16.61] | 5.20 [-6.90 to 11.90]

3. Primary Outcome: Absolute Muscle Volume Growth Rate of the Medial Gastrocnemius and the Distal Compartment of the Semitendinosus
Description: Estimation of the absolute muscle volume growth rate, calculated by: (muscle volume (mL)post-muscle volume pre)/(age (months)post-age (months)pre)
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: ml/month
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 25 | 20
ml/month
  Medial Gastrocnemius | 0.00 [-1.34 to 0.97] | 0.17 [-0.23 to 0.87]
  Semitendinosus: number analyzed (Participants) | 24 | 19
  Semitendinosus | -0.49 [-1.45 to 0.58] | 0.02 [-0.39 to 0.48]

4. Primary Outcome: Change in Kinematic Parameters
Description: Estimation of the kinematic parameters throughout the whole gait cycle by three-dimensional gait analysis.
Time Frame: Between baseline and 8-10 weeks after the BoNT injections
Population: Control group: 3DGA was not performed
Measure: Median (Inter-Quartile Range); unit: Degrees
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 25 | 0
Degrees
  Ankle Range of Motion in Sagittal Plane | -1.74 [-9.04 to 3.07] |
  Ankle Angle in Sagittal Plane at Initial Contact | 3.56 [0.47 to 6.36] |
  Maximal Ankle Angle in Sagittal Plane During Stance Phase | 3.99 [-0.32 to 9.99] |
  Maximal Ankle Angle in Sagittal Plane During Swing Phase | 5.34 [1.16 to 9.70] |
  Knee Range of Motion in Sagittal Plane | 1.94 [-3.79 to 8.84] |
  Knee Angle in Sagittal Plane at Initial Contact | -1.69 [-9.19 to 1.84] |
  Minimal Knee Angle in Sagittal Plane During Stance | -2.44 [-7.61 to 2.23] |

5. Primary Outcome: Change in Gait Profile Score (Degrees)
Description: The Gait Profile Score (GPS) is a summary measure derived from three-dimensional gait analysis that quantifies the overall deviation of a patient's gait kinematics from a normative (typically developing) reference dataset. It is calculated as the root mean square difference between the patient's joint angle trajectories of the lower limb and the corresponding mean trajectories of typically developing individuals across a gait cycle. The GPS is expressed in degrees and is based on nine key kinematic variables: pelvic tilt, obliquity, rotation; hip flexion, abduction, rotation; knee flexion; ankle dorsiflexion; and foot progression angle, typically for both left and right sides. It provides a global index of gait abnormality, where lower scores indicate gait patterns closer to normal, and higher scores reflect greater kinematic deviation.
Time Frame: Between baseline and 8-10 weeks after the BoNT injections
Population: Control group: 3DGA was not performed
Measure: Median (Inter-Quartile Range); unit: Degrees
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 25 | 0
Degrees | -1.76 [-2.51 to -0.15] |

6. Primary Outcome: Change in the Spatial-temporal Parameter "Cadence".
Description: Estimation of the cadence by three-dimensional gait analysis.
Time Frame: Between baseline and 8-10 weeks after the BoNT injections
Population: Control group: 3DGA was not performed
Measure: Median (Inter-Quartile Range); unit: Number of steps/second
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 25 | 0
Number of steps/second | -0.05 [-0.28 to 0.10] |

7. Primary Outcome: Change in the Spatial-temporal Parameter "Walking Velocity".
Description: Estimation of the walking velocity by three-dimensional gait analysis.
Time Frame: Between baseline and 8-10 weeks after the BoNT injections
Population: Control group: 3DGA was not performed
Measure: Median (Inter-Quartile Range); unit: Meter/second
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 25 | 0
Meter/second | 0.01 [-0.10 to 0.10] |

8. Primary Outcome: Change in the Spatial-temporal Parameter "Stride Length".
Description: Estimation of the stride length by three-dimensional gait analysis.
Time Frame: Between baseline and 8-10 weeks after the BoNT injections
Population: Control group: 3DGA was not performed
Measure: Median (Inter-Quartile Range); unit: Meters
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 25 | 0
Meters | 0.02 [-0.03 to 0.08] |

9. Primary Outcome: Change in Spasticity of the Medial Gastrocnemius and the Medial Hamstrings
Description: Muscle activity of the medial gastrocnemius and the medial hamstrings as recorded by surface electromyography (millivolts) during a passive stretch at high velocity of the plantar flexors and the hamstrings.
Time Frame: Between baseline and 8-10 weeks after the BoNT injections
Population: Control group: ISA was not performed n (medial hamstrings) = 13 < 14 due to insufficient cooperation
Measure: Median (Inter-Quartile Range); unit: µV
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 14 | 0
µV
  Medial Gastrocnemius | -4.73 [-15.74 to 1.31] |
  Medial Hamstrings: number analyzed (Participants) | 13 | 0
  Medial Hamstrings | -2.82 [-7.64 to 0.21] |

10. Secondary Outcome: Change in Normalized Muscle Tendon Unit Length of the Medial Gastrocnemius
Description: Estimation of the muscle tendon unit length by three-dimensional freehand ultrasonography, expressed as a percentage of total leg length.
Time Frame: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: a percentage of total leg length
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 25 | 20
a percentage of total leg length | 0.88 [-0.22 to 1.59] | -0.35 [-0.86 to 0.52]

11. Secondary Outcome: Change in Normalized Muscle Belly Length of the Medial Gastrocnemius and the Distal Compartment of the Semitendinosus
Description: Estimation of the muscle belly length by three-dimensional freehand ultrasonography, expressed as a percentage of total leg length.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: a percentage of total leg length
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 25 | 20
a percentage of total leg length
  Medial Gastrocnemius | 0.44 [0.03 to 1.25] | -0.13 [-0.92 to 0.71]
  Semitendinosus: number analyzed (Participants) | 24 | 19
  Semitendinosus | -0.32 [-0.90 to 1.47] | -0.22 [-0.74 to 0.83]

12. Secondary Outcome: Change in Normalized Tendon Length of the Medial Gastrocnemius
Description: Estimation of the tendon length by three-dimensional freehand ultrasonography, expressed as a percentage of total leg length.
Time Frame: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: a percentage of total leg length
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 25 | 20
a percentage of total leg length | -0.03 [-0.88 to 1.17] | -0.26 [-0.55 to 0.24]

13. Secondary Outcome: Normalized Muscle Volume Growth Rates of the Medial Gastrocnemius and the Distal Compartment of the Semitendinosus
Description: Estimation of the normalized muscle volume growth rates, calculated by (Normalized muscle volume (mL/kg*m)post-Normalized muscle volume pre (mL/kg*m))/(age (months)post-age (months)pre)
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: ml/kg*m/month
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 25 | 20
ml/kg*m/month
  Medial Gastrocnemius | -0.02 [-0.07 to 0.03] | 0.01 [-0.04 to 0.02]
  Semitendinosus: number analyzed (Participants) | 24 | 19
  Semitendinosus | -0.02 [-0.08 to 0.01] | -0.00 [-0.03 to 0.02]

14. Secondary Outcome: Change in the Kinematic Parameter "Ankle Range of Motion in Sagittal Plane During Stance Phase"
Description: Estimation of ankle range of motion in sagittal plane during stance phase by three-dimensional gait analysis.
Time Frame: Between baseline and 8-10 weeks after the BoNT injections
Population: Control group: 3DGA was not performed
Measure: Median (Inter-Quartile Range); unit: Degrees
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 25 | 0
Degrees | 0.31 [-4.38 to 3.74] |

15. Secondary Outcome: Change in the Kinematic Parameter "Knee Range of Motion in Sagittal Plane During Stance Phase"
Description: Estimation of knee range of motion in sagittal plane during stance phase by three-dimensional gait analysis.
Time Frame: Between baseline and 8-10 weeks after the BoNT injections
Population: Control group: 3DGA was not performed
Measure: Median (Inter-Quartile Range); unit: Degrees
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 25 | 0
Degrees | 3.68 [-0.43 to 6.91] |

16. Secondary Outcome: Change in Muscle Activation of the Medial Gastrocnemius and the Medial Hamstrings (i.e. the Change During the High-velocity Stretch).
Description: Calculated by subtracting the muscle activation during a low-velocity stretch. Muscle activity of the medial gastrocnemius and Medial Hamstrings is recorded by surface electromyography (millivolts) during a passive stretch of the plantar flexors and of the hamstrings.
Time Frame: Between baseline and 8-10 weeks after the BoNT injections
Population: Control group: ISA was not performed n (medial hamstrings) = 13 < 14 due to insufficient cooperation
Measure: Median (Inter-Quartile Range); unit: µV
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 14 | 0
µV
  Medial Gastrocnemius | -2.64 [-8.06 to 2.48] |
  Medial Hamstrings: number analyzed (Participants) | 13 | 0
  Medial Hamstrings | -3.13 [-5.78 to 0.87] |

17. Secondary Outcome: Change of Range of Motion in the Ankle and Knee Joint
Description: Evaluation by goniometry expressed in degrees. For the ankle plantar flexion range of motion with the knee extended, for the hamstrings unilateral popliteal angle.
Time Frame: Between baseline and 8-10 weeks after the BoNT injections
Population: A standardized clinical examination was performed during the pre- and post-BoNT-A assessments of the intervention group and during the pre-assessment of the control group. These data were used to describe and compare both groups at baseline.
Measure: Median (Inter-Quartile Range); unit: Degrees
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 25 | 0
Degrees
  Plantar flexors | 0.0 [0.00 to 5.0] |
  Hamstrings | 0.0 [-0.5 to 1.3] |

ADVERSE EVENTS:
Time Frame: Between baseline and 8-10 weeks after the BoNT injections for the intervention group, and between baseline and 8-10 weeks later for the control group.
Arm/Group | Intervention Group | Control Group
All-Cause Mortality (participants affected / at risk) | 0/25 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/25 | 0/20
Other Adverse Events (participants affected / at risk) | 0/25 | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-05-10): https://cdn.clinicaltrials.gov/large-docs/93/NCT05126693/Prot_SAP_000.pdf